CLINICAL TRIAL: NCT02409615
Title: A Pilot Study of the Effectiveness of Complementary Therapies to Reduce Pain in Spinal Fusion Patients
Brief Title: Complementary Therapies in Spinal Fusion Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: Healing Touch Worldwide Foundation (Other)
Responsible Party: Principal Investigator, Karen Sacks, MSN, PNP, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KS001
Record Dates: First submitted 2015-04-01; First posted 2015-04-07 (Estimated); Results first posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Idiopathic Scoliosis
Keywords: Complementary therapies; Hypnosis; Healing Touch

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Hypnosis Group (Active Comparator): Hypnosis Group: ten participants will receive Hypnosis therapy in addition to the standard postoperative pain management protocol
  Interventions: Other: Hypnosis Therapy
- Healing Touch Group (Active Comparator): Healing Touch Group: ten participants will receive Healing Touch therapy in addition to the standard postoperative pain management protocol
  Interventions: Other: Healing Touch Therapy
- Control Group (No Intervention): Control Group: ten participants will receive standard postoperative pain management protocol

INTERVENTIONS:
Other: Hypnosis Therapy — A technique called Wakeful Hypnosis that involves suggestions for healing given to a person while in a normal state of consciousness
  Arms: Hypnosis Group
Other: Healing Touch Therapy — Healing Touch An energery based therapy that uses light body or above body touch to help balance the energy field and energy centers of the body to restore harmony within the body for greater healing.
  Arms: Healing Touch Group

SUMMARY:
In this pilot study, our central hypothesis is that two CAM modalities, hypnosis and healing touch as adjunct therapies to the standard of care, will improve analgesic use for post operative pain. In this pilot study the investigators will randomize 30 adolescents undergoing spinal fusion for idiopathic scoliosis to two test groups: Hypnosis with Pain Management Standard of Care for Post Op Pain, Healing Touch with Pain Management Standard of Care, and a control group (Pain Management Standard of Care only).

DETAILED DESCRIPTION:
Female adolescents with the diagnosis of idiopathic scoliosis requiring surgery will be approached by a member of the research team at the pre-surgical evaluation visit to participate in the study. Randomization will be done at the time of the pre-surgical visit. Microsoft Excel will be used to generate a random group assignment table to one of the following groups:

CONTROL GROUP: Standard Pain Management for Idiopathic Posterior Spinal Fusion Surgery

HYPNOSIS GROUP: Standard Pain Management for Idiopathic Posterior Spinal Fusion and Hypnosis intervention consisting of induction to achieve a state of focused attention with heightened receptivity for acceptable suggestions targeting relaxation, comfort and healing.

HEALING TOUCH GROUP: Standard Pain Management for Idiopathic Posterior Spinal Fusion Surgery and Healing Touch intervention (Chakra Connection, Magnetic Clearing)

Protocol:

1. Potential patients identified by Orthopedic surgery schedule and review of electronic medical record (EMR) for eligibility.
2. Randomization of participants into group, CPASS anxiety scale and cortisol level obtained for all participants at preoperative visit.
3. Day of surgery: Hypnosis intervention or Healing Touch intervention prior to surgical procedure by research staff
4. Intra-operative procedure: Hypnosis participant will have taped Hypnosis script during surgical procedure; Healing Touch participant will receive one minute of intentional healing at designated time each hour by Healing Touch Practitioner. Cortisol level will be obtained on all participants.
5. PACU procedure: Healing Touch intervention or Hypnosis intervention by research staff.
6. POD #1 until discharge: daily Healing Touch or Hypnosis intervention by research staff
7. POD # 2: CPASS anxiety scale and cortisol level obtained on all participants
8. Post-op analgesic regimen: Morphine PCA > 50 kg (demand 1 mg, 10 minute lockout, basal rate 0.5 mg/hr) and Morphine PCA < 40-49 kg (demand 0.8 mg, 10 minute lockout, basal rate 0.4 mg/hr), benzodiazepine, gabapentin, ketorolac and clonidine per standard protocol for all participants.
9. Pain scores (self-report), vital signs, opioid consumption, side effects, day of ambulation, transition to oral analgesics will be collected from EMR until day of discharge.
10. 4-week Postoperative visit: CPASS anxiety scale, cortisol level and pill count obtained on all participants.

Methods:

Statistical Analysis: Descriptive Statistics: Standard Descriptive Statistics will be used to describe the outcomes, demographic and independent variables of interest pre- and post-intervention, overall and by intervention group. Changes in outcomes will also be calculated and descried. For continuous variables means, medians and ranges will be produced, while frequencies and percentages will be produced for categorical variables. Means, standard deviations, medians and ranges will be computed for measured continuous variables; marginal distributions will be used for categorical factors. Graphical methods including histograms, scatterplots, and boxplots, will be used in order to understand aspects of data quantity and examine assumptions (such as normality) underlying statistical models.

The primary outcome is decrease in opioid consumption as well as reported pain and anxiety scores. We will compare difference in pain pre- to post- between the two intervention and control groups, using ANOVA. Since data will be collected at multiple points pre- and post-intervention, and some randomly missing data expected, the primary analysis will employ generalized estimating equations (GEEs). The GEEs models will be adjusted for baseline characteristics, such as age, gender, race and any important clinical characteristics. GEEs will also be used to compare the changes in reported pain and analgesic use between the three groups.

ELIGIBILITY:
Inclusion Criteria:

1. Females, ages 12 - 17
2. Diagnosis of idiopathic scoliosis

Exclusion Criteria:

1. Patients with chronic or severe disease conditions requiring spinal fusion surgery.
2. Children with profound mental disabilities or developmental delay not allowing them to voluntarily assent to participate.

Ages: 12 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2014-08; Primary Completion 2017-03-27 (Actual); Study Completion 2017-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Sacks, MSN, PNP, Principal Investigator — Nemours / A I duPont Hospital for Children
Locations (1):
- Nemours / A I duPont Hospital for Children, Wilmington, Delaware, United States

REFERENCES:
- [Background] Kemper KJ, Vohra S, Walls R; Task Force on Complementary and Alternative Medicine; Provisional Section on Complementary, Holistic, and Integrative Medicine. American Academy of Pediatrics. The use of complementary and alternative medicine in pediatrics. Pediatrics. 2008 Dec;122(6):1374-86. doi: 10.1542/peds.2008-2173. PMID 19047261
- [Background] Barnes PM, Bloom B, Nahin RL. Complementary and alternative medicine use among adults and children: United States, 2007. Natl Health Stat Report. 2008 Dec 10;(12):1-23. PMID 19361005
- [Background] Sanders H, Davis MF, Duncan B, Meaney FJ, Haynes J, Barton LL. Use of complementary and alternative medical therapies among children with special health care needs in southern Arizona. Pediatrics. 2003 Mar;111(3):584-7. doi: 10.1542/peds.111.3.584. PMID 12612240
- [Background] Post-White J, Fitzgerald M, Hageness S, Sencer SF. Complementary and alternative medicine use in children with cancer and general and specialty pediatrics. J Pediatr Oncol Nurs. 2009 Jan-Feb;26(1):7-15. doi: 10.1177/1043454208323914. Epub 2008 Oct 20. PMID 18936292
- [Background] Hagen LE, Schneider R, Stephens D, Modrusan D, Feldman BM. Use of complementary and alternative medicine by pediatric rheumatology patients. Arthritis Rheum. 2003 Feb 15;49(1):3-6. doi: 10.1002/art.10931. PMID 12579587
- [Background] Lew MW, Kravits K, Garberoglio C, Williams AC. Use of preoperative hypnosis to reduce postoperative pain and anesthesia-related side effects. Int J Clin Exp Hypn. 2011 Oct-Dec;59(4):406-23. doi: 10.1080/00207144.2011.594737. PMID 21867377
- [Background] Accardi MC, Milling LS. The effectiveness of hypnosis for reducing procedure-related pain in children and adolescents: a comprehensive methodological review. J Behav Med. 2009 Aug;32(4):328-39. doi: 10.1007/s10865-009-9207-6. Epub 2009 Mar 3. PMID 19255840

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Control Group; ten participants will receive standard postoperative pain management protocol
Period: Overall Study
Arm/Group | Hypnosis Group | Healing Touch Group | Control Group
Started | 10 | 10 | 10
Completed | 10 | 9 | 10
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Healing Touch Group: Healing Touch Group: nine participants will receive Healing Touch therapy in addition to the standard postoperative pain management protocol
  Healing Touch Therapy: Healing Touch An energery based therapy that uses light body or above body touch to help balance the energy field and energy centers of the body to restore harmony within the body for greater healing.
- Total: Total of all reporting groups
Arm/Group | Hypnosis Group | Healing Touch Group | Control Group | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.1 (1.37) | 15.0 (1.7) | 13.9 (0.74) | 14.67 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 10 | 30
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Cobb Angle [Mean (Standard Deviation); unit: degrees] — The Cobb Angle is a measurement of bending disorders of the vertebral column such as scoliosis. The Cobb Angle is measured in degrees, with a range of 10-20 to be considered mild scoliosis. Surgical treatment is generally indicated for curves exceeding 45-50 degrees.
  degrees | 53.9 (7.23) | 54.9 (1.65) | 57.5 (11.64) | 55.43 (8.31)

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain (Total Opioid Use)
Description: Total Opioid use will be measured in mg/kg/hour daily until discharge, and at postoperative follow-up visit. Postoperative time in PACU starts on admission to PACU until discharged to general nursing care floors. Postoperative Day #0 (POD #0) start on the day of surgery from the time the patient is discharged from the PACU to 7:00 AM the following morning. POD #1 is from 07:00 the day after surgery to the following morning (24 hour period) at 07:00. POD #2, POD #3 are the following 24 hour periods until time of discharge. The first outpatient postoperative appointment was four weeks after surgery.
Time Frame: up to postoperative day 4
Population: opioid comsumption calculated in morphine equivalents - mg/kg/hour
Measure: Mean (95% Confidence Interval); unit: mg/kg/hr
Arm/Group | Hypnosis Group | Healing Touch Group | Control Group
Number analyzed (Participants) | 10 | 9 | 10
mg/kg/hr
  PACU opioid use | 0.041 [0.022 to 0.061] | 0.048 [0.024 to 0.072] | 0.054 [0.027 to 0.080]
  Postoperative Day 0 | 0.038 [0.029 to 0.047] | 0.042 [0.029 to 0.054] | 0.042 [0.029 to 0.054]
  Postoperative Day 1 | 0.019 [0.015 to 0.024] | 0.023 [0.016 to 0.031] | 0.021 [0.015 to 0.027]
  Postopertive Day 2 | 0.012 [0.009 to 0.016] | 0.017 [0.010 to 0.024] | 0.012 [0.009 to 0.016]
  Postoperative Day 3 | 0.012 [0.009 to 0.015] | 0.011 [0.006 to 0.017] | 0.011 [0.005 to 0.018]
  Postoperative Day 4: number analyzed (Participants) | 1 | 2 | 5
  Postoperative Day 4 | 0.02 [0.000 to 0.020] | 0.016 [-0.111 to 0.143] | 0.014 [-0.002 to 0.029]

2. Secondary Outcome: Pain Score
Description: Average pain score utilizing Visual Analog Scale which is a self report pain scale from 0 - 10 with a score of "0" indicating no report of pain and a score of "10" indicating the worst pain imaginable.
Time Frame: up to postoperative day 4
Population: One participant was withdrawn from the study. Day of discharge varied among participants
Measure: Mean (Standard Deviation); unit: numeric pain score
Arm/Group | Healing Touch Group | Hypnosis Group | Control Group
Number analyzed (Participants) | 9 | 10 | 10
numeric pain score
  Pain score - preoperative | 0.11 (0.33) | 0.5 (1.58) | 1.5 (2.27)
  Pain Score - PACU | 5.0 (2.24) | 4.7 (3.58) | 6.2 (1.98)
  Pain Score - POD #0 | 5.2 (1.97) | 5.18 (2.17) | 5.36 (2.0)
  Pain Score - POD #1 | 4.78 (1.69) | 4.70 (1.99) | 4.33 (1.73)
  Pain Score - POD #2: number analyzed (Participants) | 8 | 10 | 9
  Pain Score - POD #2 | 5.56 (1.48) | 5.0 (1.7) | 5.0 (1.3)
  Pain Score - POD #3: number analyzed (Participants) | 8 | 10 | 9
  Pain Score - POD #3 | 7.12 (1.46) | 5.8 (2.15) | 7.8 (1.64)
  Pain Score - POD #4: number analyzed (Participants) | 1 | 2 | 5
  Pain Score - POD #4 | 4.0 (0) | 5.8 (1.34) | 4.5 (3.36)

3. Secondary Outcome: Cortisol Level
Description: Cortisol levels obtained at 4 points - pre-operative surgical evaluation visit, intra-operative, POD #2, 4-week postoperative follow-up clinic visit. Cortisol is a hormone released by the adrenal glands. Cortisol mainly helps regulate the body's response to stress. For most tests, the normal ranges are: 6 a.m. to 8 a.m.: 10 to 20 micrograms per deciliter (mcg/dL). Around 4 p.m.: 3 to 10 mcg/dL. Normal ranges can vary from lab to lab, time to time and person to person.
Time Frame: up to 4-week postoperatively
Measure: Mean (Standard Deviation); unit: mcg/dL
Arm/Group | Hypnosis Group | Healing Touch Group | Control Group
Number analyzed (Participants) | 10 | 9 | 10
mcg/dL
  Preoperative coristol level | 4.36 (1.88) | 6.07 (2.39) | 5.03 (1.34)
  Intraoperative cortisol level | 2.94 (2.95) | 3.28 (3.67) | 3.25 (4.75)
  POD #2 cortisol level | 7.82 (3.71) | 3.80 (2.48) | 9.07 (11.55)
  Four week postoperative cortisol level | 6.09 (2.54) | 8.2 (3.2) | 6.05 (1.69)

4. Secondary Outcome: Child Pain Anxiety Symptoms Scale (CPASS)
Description: Child Pain Anxiety Symptoms Scale (CPASS) is a validated 20-item self-report tool measuring pain anxiety in adolescents undergoing major surgical procedures and obtained on all participants at 3 points - pre-surgical evaluation, POD #2 and 4-week postoperative follow-up visit. Total score is ranged from 0-100. CPASS scores ranging from 0 to 34 indicated mild pain anxiety; 35 to 67 indicated moderate pain anxiety; 68 to 100 indicated severe pain anxiety.
Time Frame: up to 4 weeks postoperatively
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hypnosis Group | Healing Touch Group | Control Group
Number analyzed (Participants) | 10 | 9 | 10
units on a scale
  Preoperative CPASS score | 19.6 (10.32) | 18.0 (11.44) | 30.3 (13.58)
  POD #2 CPASS score | 41.7 (23.92) | 41.33 (26.63) | 48.6 (11.39)
  Four week postoperative CPASS score | 21.1 (16.07) | 15.0 (9.72) | 36.89 (16.22)

ADVERSE EVENTS:
Time Frame: Postoperative Day #0 up to POD #1
Description: Participant assigned to Healing Touch Group, somnolent postoperative day #0, transferred to PICU for closer monitoring, withdrawn from study.
Groups:
- Healing Touch Group: Healing Touch Group: ten participants will receive Healing Touch therapy in addition to the standard postoperative pain management protocol
  Healing Touch Therapy: Healing Touch An energy based therapy that uses light body or above body touch to help balance the energy field and energy centers of the body to restore harmony within the body for greater healing.
Arm/Group | Healing Touch Group | Hypnosis Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 0/10 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healing Touch Group (N=10) | Hypnosis Group (N=10) | Control Group (N=10)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Participants
somnolence (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) — Postoperative somnolence. Participant transferred to PICU for additional monitoring. Once admitted to PICU, became ineligible and withdrawn from study
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healing Touch Group (N=10) | Hypnosis Group (N=10) | Control Group (N=10)
Somnulence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Participant becoming somnolent on standard weight based dosing of opioid medication, transferred to the PICU for closer monitoring. Withdrawn from study due to transfer to ICU.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-06-23): https://cdn.clinicaltrials.gov/large-docs/15/NCT02409615/Prot_SAP_000.pdf